CLINICAL TRIAL: NCT05600738
Title: Network Effects of Therapeutic Deep Brain Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sandipan Pati, MD, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSC-MS-22-0045
Record Dates: First submitted 2022-10-25; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Intractable Epilepsy
Keywords: Deep brain stimulation (DBS); neuromodulation therapy; Responsive Neurostimulation (RNS)
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: RNS/DBS activation

INTERVENTIONS:
Device: RNS/DBS activation — This will be performed to study the EEG responses to DBS/RNS stimulation electrical pulses. The stimulation frequencies will be sequentially increased and each stimulation will last for 2 minutes.There will be a 1-2 minute wash out period after each trial.

SUMMARY:
The purpose of this study is to map the acute, short-term cortical evoked responses to thalamic electrical stimulation in persons with intractable epilepsy

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Epilepsy
* undergoing neuromodulation therapy with clinically implanted neuromodulation devices (DBS, RNS)
* followed in the outpatient epilepsy clinic

Exclusion Criteria:

* pregnant women
* active psychosis, major depression, or suicidal ideation in the preceding year
* Intelligence quotient (IQ) less than 70 as measured by clinical neuropsychological evaluation
* Do not agree to share their medical records for research purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in amplitude of evoked potentials metrics as assessed by the scalp EEG | Baseline, Intra intervention (about 20 minutes after baseline)
Change in amplitude of evoked potentials metrics as assessed by the scalp EEG | Baseline, post intervention (about 2 hours after baseline )
Change in latencies of evoked potentials and phase synchronization metrics recorded as assessed by the scalp EEG | Baseline, Intra intervention (about 20 minutes after baseline)
Change in latencies of evoked potentials and phase synchronization metrics recorded as assessed by the scalp EEG | Baseline, post intervention (about 2 hours after baseline )

SECONDARY OUTCOMES:
Change in reaction time to visual stimuli measured as vigilance score assessed by the Psychomotor Vigilance test (PVT) | Baseline, Intra intervention (about 20 minutes after baseline)
  This is a computerized testing that will record errors in being unable to tap a switch/button
Change in reaction time to visual stimuli measured as vigilance score assessed by the Psychomotor Vigilance test (PVT) | Baseline, post intervention (about 2 hours after baseline)
  This is a computerized testing that will record errors in being unable to tap a switch/button

CONTACTS AND LOCATIONS:
Overall Officials: Sandipan Pati, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No